CLINICAL TRIAL: NCT05561049
Title: Efficacy and Safety of Daratumumab in Combination With Bortezomib, Thalidomide, and Dexamethasone Regimens in Newly Diagnosed Multiple Myeloma With Renal Dysfunction in Real-World: A Non-interventional Prospective Multicenter Observational Study
Brief Title: Efficacy and Safety of Daratumumab in Combination With Bortezomib, Thalidomide, and Dexamethasone Regimens in Newly Diagnosed Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: D-VTD-MM07
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — daratumumab; Bortezomib; Thalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Daratumumab in Combination with Bortezomib, Thalidomide, and Dexamethasone Regimens — Daratumumab in Combination with Bortezomib, Thalidomide, and Dexamethasone Regimens

SUMMARY:
This is an observational, multi-center, non-interventional study, which is designed to evaluate the safety and efficacy of daratumumab in Combination with Bortezomib, Thalidomide, and Dexamethasone (D-VTD) Regimens in NDMM patients with renal dysfunction in real-world clinical practice. The data collected in this trial are for subjects with NDMM and renal dysfunction treated with D-VTd regimen and consist of 2 treatment phases, efficacy and safety data from induction phase and consolidation phase.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed multiple myeloma;
2. age over 18 years, male or female;
3. glomerular filtration rate (eGFR) < 40 mL/min
4. Patients must have the ability to understand and voluntarily sign the informed consent form, which must be signed before any trial process;
5. patients who completed at least one course of treatment were included in the safety observation;
6. Patients who completed at least 2 courses of treatment were included in the efficacy observation;

Exclusion Criteria:

1. acute and chronic renal insufficiency not caused by myeloma;
2. are receiving any other investigational drug or investigational medical device;
3. Patients with other cancers confirmed before MM diagnosis, except cervical carcinoma in situ or scaly cell carcinoma of the skin and basal cell carcinoma that are considered cured for more than 3 years before enrollment;
4. patients who do not complete a course of DVTd treatment for any reason, unless permanent discontinuation or death due to the drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. newly diagnosed MM;
  2. age over 18 years, male or female;
  3. glomerular filtration rate (eGFR) < 40 mL/min
  4. patients who completed at least one course of treatment were included in the safety observation;
  5. Patients who completed at least 2 courses of treatment were included in the efficacy observation;
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Very good partial response (VGPR) rate | 28 days after consolidation therapy